CLINICAL TRIAL: NCT04552912
Title: Testing a Nurse-Led Evidence-Based Exercise Program to Improve Patient-Reported Outcomes in Adults With Acute Leukemia
Brief Title: Physical Activity to Improve Patient Reported Outcomes for Adults With Acute Leukemia
Acronym: Build Stamina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00106590
Record Dates: First submitted 2020-09-04; First posted 2020-09-17 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-08

CONDITIONS: Physical Activity; Exercise; Acute Leukemia; Consolidation; Maintenance Therapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Build Stamina Group (Experimental): The Build StaMINA (Biobehavioral Self-Management INtervention using physical Activity) is a tailored evidence-based physical activity (PA) program designed to improve endurance, strength, and balance which are all areas of physical function, that adults with acute leukemia (AL) post-induction are known to have diminished capacity. The Build StaMINA program will be tailored to their current Physical Function, per assessment. The detailed PA prescription includes each exercise in the program as well as the frequency, number of repetitions each day and rate of perceived exertion (RPE) for each exercise. The repetitions and RPE are based on the participants' current Physical Function Assessment and will be assigned based on our evidence-based algorithm.
  Interventions: Behavioral: Build Stamina Program
- Attention-Control Group (No Intervention): Participants assigned to the attention control group will have a Physical Function Assessment at baseline after informed consent has been provided and prior to randomization. Participants will also be asked to complete questionnaires regarding at baseline, 6-weeks and 3 months. Those in the attention-control group will also receive a newsletter detailing the benefits of participating in regular PA as well as regular phone calls by study team to discuss general health and wellbeing at the same schedule as intervention group.

INTERVENTIONS:
Behavioral: Build Stamina Program — Build StaMINA intervention is a self-management intervention that provides information, motivation, behavioral skills to engage in PA, and ultimately a tailored PA program for adults with AL who are receiving consolidation/maintenance chemotherapy.
  Arms: Build Stamina Group

SUMMARY:
The purpose of this study is to test the efficacy of an evidence-based tailored physical activity program adapted for adults with acute leukemia. Implementation-related process evaluation of the physical activity program will also be assessed.

DETAILED DESCRIPTION:
Rationale/Significance of Study: Acute leukemias (AL) are an aggressive and often debilitating cancer with increasing incidence among those with a prior history of cancer and older adults. Initial treatment is complex and even when remission is initially achieved, there is a high risk for disease relapse. Research shows that individual characteristics such as decreased physical function are associated with poor survival in AL. Intensive chemotherapy remains the standard treatment necessary for survival. Chemotherapy administration entails extended hospitalization for treatment and to monitor and manage multiple symptoms, life-threatening complications, and other adverse events which often necessitate intensive care unit admissions. Given the significance of this illness and its complications, adults with AL are commonly encouraged to rest during induction treatment. Unfortunately, the long periods of hospitalization and rest result in diminished physical function during and after treatment. In fact, patients are unable to function at pre-cancer levels which can delay or prevent future intensive treatments, such as hematopoietic stem cell transplant, that are most likely to be life-saving. Currently there are no clinical interventions specific to assisting adults recovering from intense induction treatment. However, PA programs have been shown to improve physical function and reduce symptoms in many other clinical/disease contexts. Specifically, the Otago home-based program, has undergone extensive testing internationally and has demonstrated effectiveness for improving strength, mobility, balance and preventing falls in vulnerable older adults. Efforts to assess the clinical efficacy of evidence-based PA programs for adults recovering from induction treatment for AL are critically needed.

Conceptual/Theoretical Framework: The evaluation approach for this study is guided by the RE-AIM (reach, efficacy, adoption, implementation, maintenance) evaluation framework. The tailored PA intervention is guided by the information-motivation-behavioral (IMB) change theory.

Main Research Variable(s): Reach: percent of eligible patients enrolled; Efficacy: physical function assessments; Adoption: qualitative interviews to understand what is needed to adopt the intervention into practice; Implementation: intervention fidelity/adherence; Maintenance: qualitative interviews to understand what is needed to sustain the intervention in practice.

Design: This is a two-group randomized controlled trial (RCT) with an implementation-related process evaluation of the tailored PA intervention. Participants will be randomized to either the nurse-led PA intervention or the attention-control group.

Setting: NCI designated Comprehensive Cancer Center Sample: Adults diagnosed with AL receiving consolidation/maintenance chemotherapy Methods: A longitudinal RCT over 3-months to evaluate the efficacy of our nurse-led tailored home-based PA program versus attention-control. Participants will complete physical function tests and questionnaires at baseline, 6-weeks and 3-months. Both quantitative and qualitative data will be collected for summative and formative data relevant to the reach, adoption, implementation, and maintenance domains of RE-AIM.

Implications for Practice: Adults with AL experience decreased physical function and concurrent symptoms that negatively affects quality of life (QOL) and may increase their risk for further adverse events. This intervention would provide oncology nurses with tools to support patients to engage in behaviors that improve their QOL.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Diagnosed with either acute leukemia
* Receiving either maintenance or consolidation chemotherapy
* Able to walk independently for 4 meters with or without gait aid.

Exclusion Criteria:

* non-English speaking
* receiving induction chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Physical Function- Short Physical Performance Battery Protocol | 12-weeks
  Measured via evaluation on Chair Stand Test (up to 4 points), Gait Speed Test (up to 4 points) and the 4 Test Balance Scale (up to 4 points) scores can range from 0-12 points. Higher scores = better physical function
Physical Function- 6 Minute walk test | 12-weeks
  The 6 minute walk Test measures an individuals ability to walk in meters for 6 minutes. The distance walk in meters is recorded. Higher meter = better physical function

SECONDARY OUTCOMES:
Patient-Reported Outcomes- Cognition | 12-weeks
  Measured via the Montreal Cognitive Assessment. Scores range from 0-30 with higher scores = better cognition
Patient-Reported Outcomes-Fatigue | 12-weeks
  Measured via Patient-Reported Outcomes Measurement Information System-Patient-Reported Outcomes Measurement Information System-Fatigue 8. Scores range from 8-40 with higher scores = worse fatigue
Patient-Reported Outcomes-Disturbed Sleep | 12-weeks
  Measured via Patient-Reported Outcomes Measurement Information System- Patient-Reported Outcomes Measurement Information SystemDisturbed Sleep 8b. Scores range from 8-40 with higher scores = worse disturbed sleep
Patient-Reported Outcomes-Anxiety | 12-weeks
  Measured via Patient-Reported Outcomes Measurement Information System-Patient-Reported Outcomes Measurement Information System-Anxiety-8. Scores range from 8-40 with higher scores = worse anxiety
Patient-Reported Outcomes-Depression | 12-weeks
  Measured via Patient-Reported Outcomes Measurement Information System- Depression-8. Scores range from 8-40 with higher scores = worse depression

CONTACTS AND LOCATIONS:
Overall Officials: Tara A Albrecht, PhD, ACNP-BC, ACNP-BC, ACHPN, Principal Investigator — Duke University School of Nursing
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No